CLINICAL TRIAL: NCT04172688
Title: Effect of Prebiotics on Function and Pain in Patients with Knee Osteoarthritis and Obesity
Brief Title: Effect of Prebiotics on Function and Pain in Patients with Osteoarthritis and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB17-2363
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Osteo Arthritis Knee; Obesity
Keywords: Pain; Gut microbiota; Prebiotic
MeSH Terms: conditions — Obesity; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Two 3.3g doses/day (12 kcal/dose) of maltodextrin
  Interventions: Dietary Supplement: Placebo maltodextrin
- Prebiotic (Experimental): Two 8g doses/day (12 kcal/dose) of oligofructose-enriched inulin
  Interventions: Dietary Supplement: Prebiotic oligofructose-enriched inulin

INTERVENTIONS:
Dietary Supplement: Prebiotic oligofructose-enriched inulin — Synergy1
  Arms: Prebiotic
Dietary Supplement: Placebo maltodextrin — Equicaloric dose of maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of the present study is to determine if prebiotic supplementation can, through changes in the intestinal gut microbiota, lead to improvements in knee function and physical performance and reduce knee pain in adults with obesity and idiopathic metabolic knee osteoarthritis. We hypothesize that prebiotics will reduce systemic and local (knee joint) inflammation, thus improving knee function, lower pain medication use, and enhance performance of daily life activities.

DETAILED DESCRIPTION:
Primary outcome:

1. To determine the change in knee joint function and physical performance in adults with obesity and knee osteoarthritis treated for 6 months with oligofructose-enriched inulin or placebo.

Secondary outcomes:

1. To determine the change in knee pain in adults with obesity and knee osteoarthritis treated for 6 months with oligofructose-enriched inulin or placebo.
2. To examine the change in body composition (fat mass and lean mass) in participants treated with oligofructose-enriched inulin or placebo.
3. To evaluate the change in quality of life in participants treated with oligofructose-enriched inulin or placebo.
4. To gain a mechanistic understanding of the influence of oligofructose-enriched inulin supplementation in metabolic OA through examination of gut microbiota composition and short-chain fatty acid concentrations.
5. To gain a mechanistic understanding of the influence of oligofructose-enriched inulin supplementation in metabolic OA through examination of serum inflammatory and metabolomics markers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 30-75 years of age.
* BMI greater than 30kg/m2.
* Diagnosis via x-ray of knee OA grade II and III (Kellgren and Lawrence).

Exclusion Criteria:

* Knee OA resulting from a traumatic injury.
* Previous knee surgery.
* Concomitant use of any weight loss medication, previous bariatric or other intestinal surgery
* Presence of active infection, pregnancy or lactation.
* Regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment.
* Antibiotic use within 3 months prior to enrollment
* Uncontrolled cardiovascular or respiratory disease, active malignancy, or chronic infections.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in 30 second chair stand test | Baseline and 6 months
  30 second chair stand test
Change in 40 metre fast based walk | Baseline and 6 months
  40 metre fast based walk
Change in Time up and go test | Baseline and 6 months
  Time up and go test
Change in 6 minute walk test | Baseline and 6 months
  6 minute walk test
Change in knee function | Baseline and 6 months
  Knee extensor torque isokinetic dynamometer (Biodex System3)

SECONDARY OUTCOMES:
Change in knee pain | Baseline and 6 months
  Numerical Pain Rating Scale (NPRS) for Knee Pain (0-10 scale)
Change in knee injury and osteoarthritis outcome score (KOOS) | Baseline and 6 months
  KOOS questionnaire (42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).)
Change in pain medication use | Baseline and 6 months
  Pain medication questionnaire
Change in body fat | Baseline and 6 months
  Body fat percent
Change in fecal microbiota composition | Baseline and 6 months
  Fecal microbiota
Change in fecal short chain fatty acids (SCFA) concentration | Baseline and 6 months
  Fecal SCFA
Change in serum endotoxin | Baseline and 6 months
  Serum LPS
Change in serum inflammatory marker | Baseline and 6 months
  Serum IL-6
Change in physical activity level | Baseline and 6 months
  ActiGraph Link® accelerometer
Change in quality of life ratings | Baseline and 6 months
  SF-36 Quality of Life Questionnaire
Change in serum metabolomics | Baseline and 6 months
  Serum LC-Qtof-Mass Spec metabolomics

OTHER OUTCOMES:
Change in gastrointestinal comfort | Baseline and 6 months
  Gastrointestinal Feelings Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortuna R, Wang W, Mayengbam S, Tuplin EWN, Sampsell K, Sharkey KA, Hart DA, Reimer RA. Effect of prebiotic fiber on physical function and gut microbiota in adults, mostly women, with knee osteoarthritis and obesity: a randomized controlled trial. Eur J Nutr. 2024 Sep;63(6):2149-2161. doi: 10.1007/s00394-024-03415-w. Epub 2024 May 7. PMID 38713231
- [Derived] Fortuna R, Hart DA, Sharkey KA, Schachar RA, Johnston K, Reimer RA. Effect of a prebiotic supplement on knee joint function, gut microbiota, and inflammation in adults with co-morbid obesity and knee osteoarthritis: study protocol for a randomized controlled trial. Trials. 2021 Apr 7;22(1):255. doi: 10.1186/s13063-021-05212-w. PMID 33827639